CLINICAL TRIAL: NCT04177303
Title: Gut-derived Incretin Hormones in the Pathophysiology of Type 1 Diabetes Mellitus; Effect of Metformin Treatment
Brief Title: Incretin Hormones in Type 1 Diabetes Mellitus;Effect of Metformin Treatment
Acronym: INCREDIBLE-M
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCREDIBLE-ME
Record Dates: First submitted 2019-10-30; First posted 2019-11-26 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Metformin; Incretin hormones; Inflammation; Microbiome
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Inflammation | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Pilot, mechanistic, phase 3, randomized, placebo-controlled, parallel designed, double-blinded clinical trial
Who Masked: Participant, Investigator
Masking Description: All pills will be provided as effervescent, pre-scored 1000mg tablets, so that they may easily be dichotomized.Boxes with active drug or placebo will be covered to conceal the identity of the test article. Sponsor will provide covering materials.The unblinded designee will provide the covered boxes to the blinded nurse or blinded investigator who will dispense the pills.Participants will be given study drug diaries, which they will complete during study drug intake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): Patients will continue with their standard insulin therapy and will additionally receive orally metformin 2gr/day.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Patients will continue with their standard insulin therapy and will additionally receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Participants will be randomized to metformin 2000 mg
  Arms: Metformin
Drug: Placebo — Participants will be randomized to placebo
  Arms: Placebo

SUMMARY:
Investigators aim is to conduct an RCT to study the effect of adjunct metformin treatment to insulin monotherapy in patients with type 1 diabetes, targeting the intestinal incretin secretion. The patients will be randomly allocated to metformin or placebo treatment for 4 months

DETAILED DESCRIPTION:
Compared to the large armamentarium of antidiabetic agents for Type 2 Diabetes Mellitus (T2DM), the insulinocentric therapeutic approach in Type 1 Diabetes Mellitus (T1DM) has distracted the scientific perspective from the rise of novel therapies. Insulin monotherapy has long overshadowed the overall hormonal dysregulation that demarcates T1DM . In specific, the significance of the gut-derived incretin hormones GLP-1 (glucagon-like peptide 1) and GIP (glucose-dependent insulinotropic peptide), which are implicated with glucose metabolism via the gut-pancreatic axis, has been merely addressed.

Investigators' goal in the current protocol is to delineate the glucoregulatory role of incretin hormones in T1DM and the therapeutic advantages of adjunct metformin treatment over insulin monotherapy. In the absence of such knowledge, the development of effective strategies to improve metabolic homeostasis and ameliorate complications in T1DM patients will remain problematic. The central hypothesis of the study is that metformin, as an incretin-secretagogue, will enhance postprandial incretin secretion in T1DM patients, which will be reflected in reduced glucagon secretion and improvement in glycemic volatility. Mechanistic insight will be provided through changes in specific amino acids and metabolites patterns, chronic inflammation and the microbiome composition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* T1DM (Diagnosis of diabetes before the age of 35 years and insulin use within 1 year of diagnosis)
* Treatment with multiple daily insulin injections (MDI) or continuous subcutaneous insulin infusion (CSII)

Exclusion Criteria:

* Any cardiovascular disease within the last 3 months
* NYHA stage 3 or 4 heart failure
* Uncontrolled angina
* Liver failure [AST>135 IU/L or ALT>129IU/L (3 x the upper normal limit)] • Kidney failure or GFR<60 ml/min/1.73m2
* Gastrointestinal disease or gastroparesis
* Prior diagnosis of cancer within 2 years
* Other medication that affect glucose metabolism within the last 3 months (metformin, SGLT2, GLP-1 analogues, amylin analogues, systemic glucocorticosteroids)
* Untreated or uncontrolled thyroid disease
* Pregnancy or breastfeeding
* Alcohol consumption > 2-drinks per day or other substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2022-11-29 (Estimated); Study Completion 2022-11-29 (Estimated)

PRIMARY OUTCOMES:
Change in GLP-1 (glucagon like peptide) and GIP (gastric inhibitory peptide) postprandial secretion | 4 months
  The primary endpoint of the study is the change in postprandial GLP-1(ng/ml) and GIP (ng/ml) secretion with metformin treatment compared to placebo.

SECONDARY OUTCOMES:
Change in glycemic variability pre- and post- treatment | 4 months
  A continuous glucose-monitoring device will be attached to each participant and record daily glucose measurements (mg/dl) for 6 consecutive days on two separate time points: a) within a week prior to randomization and b) as a follow up, within a week prior to Inpatient Visit 2.
Metabolomic profile of each treatment group | 4 months
  Untargeted metabolomics analysis and identification of candidate metabolites using mass spectrometry. Quantitative targeted metabolomics will then be applied on candidate metabolites to compare differences pre and post treatment between metformin and placebo treatment arm
Change in inflammatory state | 4 months
  Corrrelation of CRP levels (mg/dl) and treatment arm, as marker of inflammation. CRP will be measured from plasma blood samples collected during Inpatient Visits 1 and 2.
Change in endothelial dysfunction | 4 months
  Correlation of Serpin E1/PAI-1 levels (ng/ml), VEGF levels (pg/ml), ICAM1 levels (ng/ml) SYndecan-1 levels (ng/ml) and placebo/metformin administration, as markers of endothelial dysfunction. Concentration of adhesion molecules will be measured and compared from plasma blood samples collected during Inpatient Visits 1 and 2.
Change in cytokine production | 4 months
  Correlation of TNFα levels (pg/ml) ,IL-6 levels (pg/ml),IL-1β levels (pg/ml),IL-10 levels ,(pg/ml) and placebo/metformin administration, as markers of inflammation. Concentration of cytokines will be measured and compared from plasma blood samples collected during Inpatient Visits 1 and 2.
Change in matrix metalloproteinase-9 (MMP-9) levels | 4 months
  Correlation of MMP-9 levels (ng/ml) levels and placebo/metformin administration, as markers of inflammation. Concentration of MMP-9 will be measured and compared from plasma blood samples collected during Inpatient Visits 1 and 2.
Change in chemokine production | 4 months
  Correlation of CCL2 levels (pg/ml) ,CCL3 levels (pg/ml),CCL4 levels (pg/ml) and placebo/metformin administration, as markers of inflammation. Concentration chemokines will be measured and compared from plasma blood samples collected during Inpatient Visits 1 and 2.
Change in gene expression | 4 months
  RNA from PBMCs collected pre and post intervention will be isolated and Quantitative Real Time PCR will be used to measure the transcription of genes related to inflammation and endothelial function.
Change in gut microbiome analysis | 4 months
  Stool samples will be collected pre and post the intervention on Inpatient Visits 1 and 2 to identify the changes in the microbiome composition based on phylogenetic analysis of the 16S rRNA gene sequencing classification using quantitative PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Kotsa Kalliopi, MD,PhD, Principal Investigator — 1st Internal Medicine Department, AHEPA University Hospital
Locations (1):
- Diabetes Center, 1st Internal Medicine Department, AHEPA University General Hospital of Thessaloniki, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No